CLINICAL TRIAL: NCT05477940
Title: Exploratory Study on the Safety and Effectiveness of Absorbable Zinc Alloy Drug-eluting Coronary Stent System
Brief Title: Study on Absorbable Zinc Alloy Drug Eluting Coronary Stent System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Collaborators: Shandong Rientech Medical Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-R-1
Record Dates: First submitted 2022-04-26; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Coronary Heart Disease; Drug Eluting Stent
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Absorbable zinc alloy drug eluting stent system (Experimental): 1. Balloon pre dilation is required.
  2. Inject nitroglycerin, perform angiography after stent implantation, and record the specification and model of the instrument.
  3. After stent expansion, it should reach 100% - 110% of the vessel diameter, and the visual residual stenosis should be less than 20%.
  Interventions: Device: Absorbable zinc alloy drug eluting coronary stent system

INTERVENTIONS:
Device: Absorbable zinc alloy drug eluting coronary stent system — Absorbable zinc alloy drug eluting coronary stent system" (hereinafter referred to as "stent system") consists of "delivery system" and "drug stent (hereinafter referred to as stent)" pressed on the balloon end of the delivery system

SUMMARY:
This trial is a prospective, two center single group registration pilot trial aiming to evaluate the product safety, and provide information for the later confirmatory test design according to the results.

DETAILED DESCRIPTION:
This trial is a prospective, two center single group registration pilot trial with late lumen loss in stent (LLL), mace event and target lesion failure (TLF) as the main endpoint. Subjects were followed up clinically or by telephone at 1 month, 3 months, 6 months, 9 months and 12 months, and coronary angiography was performed at the target lesion segments for 6 months to calculate lumen loss. Analyze and evaluate the collected data, preliminarily evaluate the product safety, and provide information for the later confirmatory test design according to the results.

ELIGIBILITY:
Inclusion Criteria:

* (1) General inclusion criteria

  * The patient must be 18-75 years old; ② The patient has evidence of ischemia (such as chest pain or functional examination such as stress test, which determines that he has stable or unstable angina pectoris or asymptomatic myocardial ischemia) and is suitable for elective PCI;

    * The patient must be a qualified candidate for PCI; ④ Female patients of childbearing age had no pregnancy plan for up to one year after the starting operation. Women of childbearing age must have a pregnancy test and get negative results according to the regulations of the local test center 14 days before the starting operation.

      * Female patients were not breast-feeding during the screening visit and had no breast-feeding plan for up to 1 year after the starting operation; ⑥ The patient agrees not to participate in other clinical trials until the end point of this trial is reached; ⑦ The patient / legally authorized representative understands the purpose and procedure of the test and voluntarily signs the informed consent form;

Exclusion Criteria:

* ① Cardiogenic shock;

  * It is known that the left ventricular ejection fraction (LVEF) measured by quantitative analysis is less than 30%. For patients with stable coronary heart disease, LVEF measured within 6 months before operation is effective. For patients with acute coronary syndrome (ACS), LVEF must be measured before randomization to determine whether the patients meet the conditions;

    * The patient has a high risk of bleeding, or has a history of bleeding tendency and coagulation disorder; Major gastrointestinal bleeding within 6 months; Severe hematuria; There are contraindications to antiplatelet preparation and anticoagulant treatment, and antithrombotic treatment cannot be carried out;

      * Patients have allergic / hypersensitive reactions to aspirin, clopidogrel, heparin and ticlopidine hydrochloride (platelet inhibitor);

        * Patients have allergies or contraindications that inhibit the device materials and degradation products (rapamycin, polyglycolide and lactide) and cannot be completely cured before treatment.

          * The patient is allergic to contrast medium and cannot be completely cured before treatment.

            * Any surgical treatment requiring general anesthesia or interruption of aspirin or P2Y12 inhibitors is planned within 365 days after operation.

              * The patient received target vessel PCI within 365 days before operation. If the patient has received non target vessel PCI Treatment > 30 days before operation, the patient can still be enrolled in this trial.

                * Patients expected to require staged PCI of target vessels.

                  * Acute myocardial infarction within one week; A series of clinical symptoms of the patient are consistent with new acute myocardial infarction (AMI).

                    * During screening, the patient was determined to have arrhythmia according to any of the following criteria; Patient a needs coumarin or any other long-term oral anticoagulant; B patient may have hemodynamic instability due to arrhythmia; Patients with C had poor survival and prognosis due to arrhythmia;

                      * The patient had severe peripheral vascular disease and could not be safely inserted with 6F sheath;

                        * Stroke (CVA) or transient ischemic attack (TIA) occurred in the past 6 months; Intracranial hemorrhage, permanent neurological deficit, or any known intracranial lesions (such as aneurysms, arteriovenous malformations, etc.) have occurred in the past

                          ⑭ Major surgery within six weeks;

                          ⑮ Leukocyte count < 4.0 * 109cells / L and platelet count < 100 * 109cells / L;

                          ⑯ Severe renal and liver dysfunction;

                          ⑰ The life expectancy of patients is less than 12 months;

                          ⑱ The patient is receiving immunosuppressive therapy or is known to have immunosuppressive or autoimmune diseases (such as human immunodeficiency virus infection, systemic lupus erythematosus, etc.); Note: immunotherapy does not include hormone therapy;

                          ⑲ Patients who participate in clinical trials of other drugs or devices and fail to reach the main end point of the study;

                          ⑳ Patients who are unable or unwilling to participate in this trial, and the researchers believe that they are not suitable to participate in this trial.

8.2 angiographic exclusion criteria

1. The target lesion is located in the left main trunk and more than one lesion (not a single target lesion);
2. The% ds of visual or quantitative evaluation of target lesions is less than 50%, and the blood flow TIMI is less than grade 1.
3. The Dmax of target lesions measured by online QCA exceeds the range of 2.5mm-3.53.5mm, or the RVD measured by visual inspection exceeds the range of 2.5mm-3.53.5mm.
4. The visual length of target lesion or the length measured by online QCA is not within the range of ≤ 28 ≤ 28mm.
5. The target lesion of the right coronary artery (RCA) at the aortic opening (within 3mm of the aortic junction of RCA);
6. The target lesion is located within 3mm from the starting point of left anterior descending artery (LAD) or left circumflex artery (LCX).
7. The target lesion involves bifurcation and has the following characteristics:

   A side branch diameter ≥ 2mm; B diameter stenosis ≥ 50%; The C lateral branch needs to use protective guide wire or the lateral branch needs to be pre expanded.
8. Anatomical structures near or within the target lesion hinder the delivery of zinc alloy stents, including:

   A extreme reverse arch (≥ 90 °) at the proximal end of the target lesion or within the lesion; B. excessive bending of the proximal end of the target lesion or within the lesion (≥ two 45 ° angles); C moderate or severe calcification near or inside the target lesion.
9. The target lesion or target vessel involves myocardial bridge;
10. Angiographic images showed that the target vessel contained thrombus;
11. Before the starting operation, the target vessel has been treated with stent, and the zinc alloy stent will need to pass through the stent to reach the target lesion;
12. The target vessel has been treated with stent, and the target lesion is located within 5mm of the proximal end of the treated lesion;
13. The pre dilated balloon could not expand completely at the target lesion. Full expansion is based on the following criteria:

A. the stenosis rate (% DS) of participating lesion diameter must be < 40% (visual inspection); B blood flow reaches timi3 (visual inspection); C no angiographic complications (e.g. distal embolization, collateral occlusion); D no interlayer, NHLBI grade, d-f type; E no persistent chest pain (> 5 minutes) and no ST segment depression or elevation lasting > 5 minutes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
late lumen loss | 6 months after operation
  Difference between the minimum lumen diameter immediately after operation and the minimum lumen diameter 6 months after operation
incidence of target lumen failure(TLF) | 6 months after operation
  proportion of the number of patients with cardiac death, target vessel myocardial infarction, or clinical symptom driven target vessel revascularization in the total number
incidence of major adverse cardiac events(MACE) | 6 months after operation
  proportion of the number of patients with cardiac death, myocardial infarction or target lesion revascularization (TLR) in the total number
incidence of target lumen failure(TLF) | 1 months after operation
  proportion of the number of patients with cardiac death, target vessel myocardial infarction, or clinical symptom driven target vessel revascularization in the total number
incidence of major adverse cardiac events(MACE) | 1 months after operation
  proportion of the number of patients with cardiac death, myocardial infarction or target lesion revascularization (TLR) in the total number

SECONDARY OUTCOMES:
Device success rate | in the operation
  It means that the instrument can be successfully delivered to the target lesion as expected, the stent can be expanded normally, and the catheter can be successfully withdrawn to the outside of the body.
Operation Success Rate | 0 to 24 hours after intervention
  After stent implantation, stent diameter stenosis < 30% (visual), TIMI flow class 3, and hospitalization MACE events did not happen
Thrombotic events incidence | 1, 3, 6, 9 and 12 months after operation
  According to ARC definition it includes deterministic thrombosis, possible thrombosis and not eliminating thrombosis; point-in-time include acute within 24h, subacute between 2 and 30 d and later period over 30 d
incidence of target lumen failure(TLF) | 3, 9,12 months after operation
  proportion of the number of patients with cardiac death, target vessel myocardial infarction, or clinical symptom driven target vessel revascularization in the total number
incidence of major adverse cardiac events(MACE) | 3, 9,12 months after operation
  proportion of the number of patients with cardiac death, myocardial infarction or target lesion revascularization (TLR) in the total number

IPD SHARING:
Plan to Share IPD: No